CLINICAL TRIAL: NCT02115438
Title: A Cohort Study for Occupational Stress Induced Early Embryonic Death
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Yiming Zhao, Director of Research Center of Clinical Epidemiology, Peking University Third Hospital
Other Study IDs: 54416-01
Record Dates: First submitted 2014-04-14; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Etiology; Cohort Study; Early Embryonic Death; Occupational Stress; Occupational Epidemiology
MeSH Terms: conditions — Embryo Loss; Occupational Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Occupational Stress

SUMMARY:
Occupation stress can be the risk factors of early embryonic death

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women and their spouses in the gynecology clinic patients and wish to create the cards in the hospital;
2. the gestational age is less than 14 weeks;
3. pregnant women and their spouses have jobs before treatment.

Exclusion Criteria:

Do not sign the informed consent.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: pregnant women with job
Sampling Method: Non-Probability Sample
Enrollment: 3405 (Actual)
Dates: Start 2010-03; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
early embryonic death | 20 weeks